CLINICAL TRIAL: NCT07331753
Title: The Outcomes of Fat Grafting Combined With Latissimus Dorsi Muscle Flap for Delayed Breast Reconstruction After Mastectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Diaa eldeen abd elraheem mohamed, Assistant lecturer of plastic surgery sohag university, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med--25-12-2MD
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Breast Reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Female patients with breast cancer undergoing mastectomy (Active Comparator): Delayed breast reconstruction after breast cancer mastectomy
  Interventions: Procedure: Fat grafting combined with latissimus dorsi muscle flap

INTERVENTIONS:
Procedure: Fat grafting combined with latissimus dorsi muscle flap — Fat grafting combined with latissimus dorsi muscle flap for delayed breast reconstruction

SUMMARY:
The outcomes of fat grafting combined with latissimus dorsi muscle flap for delayed breast reconstruction after mastectomy

DETAILED DESCRIPTION:
The outcomes of fat grafting combined with latissimus dorsi muscle flap for delayed breast reconstruction after mastectomy

ELIGIBILITY:
Inclusion Criteria:

* female patient indicated for skin sparying mastectomy

Exclusion Criteria:

* female patients with stage 4 breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Wound infection or dehesiens | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Sohag Governorate, Egypt